CLINICAL TRIAL: NCT03670342
Title: Pilot Study of Somatostatin Receptor Imaging in Nasopharyngeal Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Singapore General Hospital (Other); A*Star (Other)
Responsible Party: Sponsor
Other Study IDs: NPC SSTR
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypothesis: To estimate the proportion of locally advanced, recurrent or metastatic nasopharyngeal cancer patients which show high somatostatin receptor density (SUVmax >10) on Ga-68 DOTATATE imaging.

Galium-68 DOTATATE: PET imaging will be performed with a PET/CT scanner. Galium-68 DOTATATE will be injected intravenously. Scanning will be performed approximately 60 minutes after the injection.

The standardized uptake value (SUV) will be used in the interpretation of the Ga-68 DOTATATE scans. The values gathered will be used as an estimate of the somatostatin receptor density. A patient will be considered to have an overall high somatostatin receptor density if the average SUVmax of all the representative lesions is more than 10.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced NPC or Metastatic NPC or locally recurrent NPC
* >21 years old
* Histological confirmation of NPC

Exclusion Criteria:

* <21 years old
* Pregnancy or breast feeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients would have to have histologically confirmed nasopharyngeal cancer and are above 21 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Number of NPC patients with high somatostatin receptor density | 60 minutes
  High somatostatin receptor density is when average maximum standardized uptake value (SUVmax) of all the representative lesions is more than 10 on Ga-68 DOTATATE imaging

CONTACTS AND LOCATIONS:
Overall Officials: Wen Long Nei, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nei WL, Jain A, Wang FQ, Khor LK, Yeong JP, Han ST, Sommat K, Ang MK, Soong YL, Loke KSH. Somatostatin receptor imaging in nasopharyngeal cancer. Ann Nasopharynx Cancer 2018;2:2
- [Derived] Lechner M, Schartinger VH, Steele CD, Nei WL, Ooft ML, Schreiber LM, Pipinikas CP, Chung GT, Chan YY, Wu F, To KF, Tsang CM, Pearce W, Morelli D, Philpott M, Masterson L, Nibhani R, Wells G, Bell CG, Koller J, Delecluse S, Yip YL, Liu J, Forde CT, Forster MD, Jay A, Dudas J, Krapp A, Wan S, Uprimny C, Sprung S, Haybaeck J, Fenton TR, Chester K, Thirlwell C, Royle G, Marafioti T, Gupta R, Indrasari SR, Herdini C, Slim MAM, Indrawati I, Sutton L, Fles R, Tan B, Yeong J, Jain A, Han S, Wang H, Loke KSH, He W, Xu R, Jin H, Cheng Z, Howard D, Hwang PH, Le QT, Tay JK, West RB, Tsao SW, Meyer T, Riechelmann H, Oppermann U, Delecluse HJ, Willems SM, Chua MLK, Busson P, Lo KW, Wollmann G, Pillay N, Vanhaesebroeck B, Lund VJ. Somatostatin receptor 2 expression in nasopharyngeal cancer is induced by Epstein Barr virus infection: impact on prognosis, imaging and therapy. Nat Commun. 2021 Jan 5;12(1):117. doi: 10.1038/s41467-020-20308-8. PMID 33402692
- See also: Somatostatin receptor imaging in nasopharyngeal cancer — http://anpc.amegroups.com/article/view/3984/4690